CLINICAL TRIAL: NCT01810588
Title: A Prospective Study of Optimal Cord Selection for Haplo-Cord Transplantation: Targeting the Inherited Paternal Antigen (IPA) and Matching for the Non-Inherited Maternal Antigen (NIMA)
Brief Title: Targeting the IPA and Matching for the Non-Inherited Maternal Antigen for Haplo-Cord Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1205012383
Record Dates: First submitted 2013-01-07; First posted 2013-03-13 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hematologic Malignancies
Keywords: Allogeneic transplant; Hematologic Malignancies; Acute Leukemia; Myeloproliferative disorders; Lymphoma; Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Myeloproliferative Disorders; Lymphoma; Neoplasms, Plasma Cell | interventions — fludarabine; fludarabine phosphate; Melphalan; Antilymphocyte Serum; thymoglobulin; Rituximab; Whole-Body Irradiation; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg (Experimental): All subjects in this cohort will receive a minimal cell dose of 2 x 10^7 total nucleated cells (TNC)/kilogram (kg) for the umbilical cord blood unit.
  Haplo-cord transplantation:
  All subjects will receive a conditioning regimen of chemotherapy prior to stem cell transplantation. No experimental drugs are used in this study, and the combinations of drugs that will be used in the conditioning regimen are combinations that have been used in the past.
  For the transplant component of treatment, subject will receive umbilical cord blood. The study involves transplantation of unlicensed units of cord blood. Therefore, these are considered investigational products.
  In addition to the umbilical cord blood unit, recipients will receive stem cells from a family member ( a haplo-identical donor). After collection and prior to infusion, these cells will be purified using a device called a CliniMACS CD34 selection device.
  Interventions: Device: CliniMACS® CD34 Reagent System; Drug: Fludarabine; Drug: Melphalan; Drug: anti-thymocyte globulin (rabbit); Drug: Rituximab; Radiation: Total Body Irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus
- Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg (Experimental): All subjects in this cohort will receive a minimal cell dose of 1 x 10^7 total nucleated cells (TNC)/kilogram (kg) for the umbilical cord blood unit.
  Haplo-cord transplantation:
  All subjects will receive a conditioning regimen of chemotherapy prior to stem cell transplantation. No experimental drugs are used in this study, and the combinations of drugs that will be used in the conditioning regimen are combinations that have been used in the past.
  For the transplant component of treatment, subject will receive umbilical cord blood. The study involves transplantation of unlicensed units of cord blood. Therefore, these are considered investigational products.
  In addition to the umbilical cord blood unit, recipients will receive stem cells from a family member ( a haplo-identical donor). After collection and prior to infusion, these cells will be purified using a device called a CliniMACS CD34 selection device.
  Interventions: Device: CliniMACS® CD34 Reagent System; Drug: Fludarabine; Drug: Melphalan; Drug: anti-thymocyte globulin (rabbit); Drug: Rituximab; Radiation: Total Body Irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus
- Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg (Experimental): All subjects in this cohort will receive a minimal cell dose of 0.5 x 10^7 total nucleated cells (TNC)/kilogram (kg) for the umbilical cord blood unit.
  Haplo-cord transplantation:
  All subjects will receive a conditioning regimen of chemotherapy prior to stem cell transplantation. No experimental drugs are used in this study, and the combinations of drugs that will be used in the conditioning regimen are combinations that have been used in the past.
  For the transplant component of treatment, subject will receive umbilical cord blood. The study involves transplantation of unlicensed units of cord blood. Therefore, these are considered investigational products.
  In addition to the umbilical cord blood unit, recipients will receive stem cells from a family member ( a haplo-identical donor). After collection and prior to infusion, these cells will be purified using a device called a CliniMACS CD34 selection device.
  Interventions: Device: CliniMACS® CD34 Reagent System; Drug: Fludarabine; Drug: Melphalan; Drug: anti-thymocyte globulin (rabbit); Drug: Rituximab; Radiation: Total Body Irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus
- Cohort 4 (Experimental): All subjects in this cohort will receive the minimum required cell dose that is determined following the dose de-escalation portion of the study (cohorts 1 through 3)
  Haplo-cord transplantation:
  All subjects will receive a conditioning regimen of chemotherapy prior to stem cell transplantation. No experimental drugs are used in this study, and the combinations of drugs that will be used in the conditioning regimen are combinations that have been used in the past.
  For the transplant component of treatment, subject will receive umbilical cord blood. The study involves transplantation of unlicensed units of cord blood. Therefore, these are considered investigational products.
  In addition to the umbilical cord blood unit, recipients will receive stem cells from a family member ( a haplo-identical donor). After collection and prior to infusion, these cells will be purified using a device called a CliniMACS CD34 selection device.
  Interventions: Device: CliniMACS® CD34 Reagent System; Drug: Fludarabine; Drug: Melphalan; Drug: anti-thymocyte globulin (rabbit); Drug: Rituximab; Radiation: Total Body Irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Device: CliniMACS® CD34 Reagent System — The stem cells from the haplo-identical donor will be purified by a procedure called CD34 selection before they are given to the subject. A special device called the CliniMACS® CD34 Reagent System, which is not FDA approved, will be used for this purpose. The manufacturer of the device, Miltenyi Biotec, is providing the researchers access to the device for use in this research study. Because the stem cells from the haplo-identical donor are treated using the CliniMACS CD34 selection device, they cells are considered investigational.
Drug: Fludarabine — Administer 30 mg/m2 /day intravenously x 5 days (Day -7 to Day -3) of a total dose of 150 mg/m2. Fludarabine will be dosed according to actual body weight.
  Other Names: Fludara, Fludarabine phosphate
Drug: Melphalan — Administer 70mg/m2/day intravenously x 2 days. Melphalan will be dosed according to actual body weight. Cryotherapy with ice chips will be administered to prevent mucositis
Drug: anti-thymocyte globulin (rabbit) — Administer 1.5 mg/kg/day intravenously x 3 days, total 4.5 mg/kg. ATG will be dosed according to actual body weight. The first dose will be infused over at least six hours, and subsequent doses over at least 4 hours. Pre-medications include acetaminophen 650 mg by mouth, diphenhydramine 25-50 mg by mouth or intravenously, and methylprednisolone 2 mg/kg (1 mg/ kg at the initiation and 1 mg/kg half-way through anti-thymocyte globulin administration).
  Other Names: rATG, Rabbit ATG
Drug: Rituximab — Administer one dose of 375 mg/m2 prior to or upon admission for all patients not previously exposed to rituximab or who have not received rituximab in the six months prior to transplant.
  Other Names: Rituxan
Radiation: Total Body Irradiation — Patients at high risk of CNS relapse (e.g. ALL or Burkitt's lymphoma) or patients at high risk for graft rejection (i.e., donor-specific HLA antibodies, patients with severe aplastic anemia, or hemoglobinopathies) may receive 2 doses of TBI as part of the conditioning.
  Other Names: TBI
Drug: Mycophenolate Mofetil — Will be started on Day -2 and given at a dose of 1000 mg every 8 hours until Day 28. Mycophenolae Mofetil can be given orally or intravenously. Infection, toxicity, very low patient weight (<50 kilograms) may prompt earlier discontinuation or adjustment of doses.
  Other Names: Cellcept, MMF
Drug: Tacrolimus — Administered 0.03/mg/kg/day intravenous continious infusion (CI) over 24 hours from 4pm Day -2 until engraftment or when subject is able to take orally, then tacrolimus approximately 0.09 mg/kg orally in 2 divided doses. Tacrolimus should be given at full dose to maintain levels of 5-15 ng/mL through Day 180, tapered by 20% every week thereafter. Infection, toxicity or other clinical circumstances may prompt earlier discontinuation or adjustment of doses. In the presence of Graft versus Host Disease, a clinical decision by the attending physician will determine if tacrolimus can be tapered or should be continued. Oral tacrolimus can be used when intravenous access for CI tacrolimus is unavailable.
  Other Names: Prograf

SUMMARY:
In this trial, we aim to improve the outcomes of haplo cord transplant. Haplo cord transplant is a novel and promising way to improve transplant outcomes. We hypothesize that identification of a graft that is at least 5/6 matched and inherited paternal antigen (IPA) targeted (i.e., cord blood grafts share one or more IPA antigens with the prospective recipient) is more important to the outcome of haplo cord transplant than the nucleated cell dose. The identification of such a graft for a large proportion of the subjects may necessitate accepting a lower umbilical cord graft dose.

In addition to a umbilical cord blood transplant, recipients will receive stem cells from a family member ( a haplo-identical donor) . After collection and prior to infusion, these cells will be purified using a device called a CliniMACS CD34 selection device. The subject will undergo a chemotherapy conditioning regimen prior to transplantation. No experimental drugs are used in this study, and the combinations of drugs that will be used in the conditioning regimen are combinations that have been used in the past.

DETAILED DESCRIPTION:
This is a clinical trial for subjects with hematologic malignancies ( acute leukemia, myeloproliferative disorders, lymphoma, myeloma) who are in need of a donor stem cell transplant, and for whom an umbilical cord blood transplant is thought to be the best option. As donors for allogeneic transplant, we typically try to use related family members, such as brothers or sisters, or volunteer donors who are 'HLA matched', i.e. share similar proteins on their cells. This study is for subjects for whom such a matched sibling donor or a matched unrelated donor is not available.

For such subjects a commonly used transplant procedure is to use stem cells from one or two umbilical cords (UCB) from a newborn. These umbilical cord blood grafts, despite not completely matching the recipient, cause few problems with graft vs host disease (a common complication of transplant). But they tend to grow very slowly and subjects often have very prolonged hospital stays and are at high risk for complications due to low blood counts. Umbilical cord blood transplant will be the standard arm for this protocol.

This study uses a new method of bone marrow transplantation called combined haplo-identical cord (haplo-cord) transplantation. In this procedure, cells from a related donor who shares half of the HLA proteins ( haplo-identical) are collected from the blood, as well as cells from an umbilical cord, and then both are transplanted. It is hoped that by using cells from a haplo-identical relative, subjects will have a faster recovery and require fewer transfusions. Over time the haplo-identical cells from the relative are replaced by the cells from the cord blood. The combined transplantation of haplo-identical stem cells and cord blood has previously been used in approximately 60 subjects with very encouraging results.

Traditionally it has been felt that the most important determinant of outcome of an UCB stem cell transplant is the cord blood cell dose. The second determinant is the degree of matching between donor and recipient. Many times, we have difficulty identifying UCB units of sufficient cell dose that are well matched. Of interest,in our prior study of haplo-cord SCT indicated outcomes seemed independent of the UCB cell dose. If this preliminary observation is correct, we may be able to improve the outcomes of haplo cord transplant further by accepting lower threshold UCB doses and rather focusing on optimal matching (including matching for HLA and another characteristic called IPA). This is the primary objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a confirmed diagnosis of:

  1. Previously Relapsed or refractory acute leukemia (myeloid or lymphoid)
  2. Acute leukemia in first remission at high-risk for recurrence
  3. Chronic myelogenous leukemia in chronic, accelerated phase or blast-crisis
  4. Recurrent or refractory malignant lymphoma or Hodgkin lymphoma
  5. Chronic lymphocytic leukemia, relapsed or with poor prognostic features
  6. Multiple myeloma
  7. Myelodysplastic syndrome
  8. Chronic myeloproliferative disease
  9. Hemoglobinopathies
  10. Aplastic anemia
  11. Other hematological disorder in need of allogeneic transplant (e.g. blastoid dendritic cell neoplasm)
* Age ≥ 18 years
* Likely to benefit from allogeneic transplant in the opinion of the transplant physician
* An HLA-identical related or unrelated donor cannot be identified within an appropriate time frame.
* Karnofsky (KPS) Performance status of >= 70%
* Acceptable organ function as defined below: Serum bilirubin: < 2.0mg/dL ALT(SGPT): < 3 X upper limit of normal Creatinine Clearance: > 50 mL/min/1.73m2 (as estimated by the modified MDRD equation)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Life expectancy is severely limited by concomitant illness or uncontrolled infection
* Severely decreased Left Ventricular Ejection Fraction (LVEF) or impaired pulmonary function tests (PFT's)
* Evidence of chronic active hepatitis or cirrhosis
* Uncontrolled HIV disease
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2028-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Gomez Arteaga, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York

REFERENCES:
- [Derived] van Besien K, Artz A, Champlin RE, Guarneri D, Bishop MR, Chen J, Gergis U, Shore T, Liu H, Rondon G, Mayer SA, Srour SA, Stock W, Ciurea SO. Haploidentical vs haplo-cord transplant in adults under 60 years receiving fludarabine and melphalan conditioning. Blood Adv. 2019 Jun 25;3(12):1858-1867. doi: 10.1182/bloodadvances.2019000200. PMID 31217161
- [Derived] van Besien K, Hari P, Zhang MJ, Liu HT, Stock W, Godley L, Odenike O, Larson R, Bishop M, Wickrema A, Gergis U, Mayer S, Shore T, Tsai S, Rhodes J, Cushing MM, Korman S, Artz A. Reduced intensity haplo plus single cord transplant compared to double cord transplant: improved engraftment and graft-versus-host disease-free, relapse-free survival. Haematologica. 2016 May;101(5):634-43. doi: 10.3324/haematol.2015.138594. Epub 2016 Feb 11. PMID 26869630

RESULTS

PARTICIPANT FLOW:
Period: Cohort 1 - Minimum Cell Dose 2 x 10^7 TN
Arm/Group | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg | Cohort 4
Started | 15 | 0 | 0 | 0
Completed | 15 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2 - Minimum Cell Dose 1 x 10^7 TN
Arm/Group | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg | Cohort 4
Started | 0 | 20 | 0 | 0
Completed | 0 | 20 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3 - Minimum Cell Dose 0.5 x 10^7
Arm/Group | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg | Cohort 4
Started | 0 | 0 | 25 | 0
Completed | 0 | 0 | 25 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 4
Arm/Group | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg | Cohort 4
Started | 0 | 0 | 0 | 210
Completed | 0 | 0 | 0 | 210
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg | Cohort 4 | Total
Number analyzed (Participants) | 15 | 20 | 25 | 210 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 15 | 164 | 203
  >=65 years | 4 | 7 | 10 | 46 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 11 | 94 | 119
  Male | 8 | 13 | 14 | 116 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 16 | 20
  Not Hispanic or Latino | 8 | 14 | 13 | 124 | 159
  Unknown or Not Reported | 7 | 5 | 9 | 70 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 30 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 4 | 2 | 2 | 37 | 45
  White | 7 | 11 | 9 | 79 | 106
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 11 | 64 | 84
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 20 | 25 | 210 | 270
Primary Disease [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia | 9 | 10 | 16 | 109 | 144
  Acute Lymphoblastic Leukemia | 1 | 3 | 2 | 17 | 23
  Chronic Myelogenous Leukemia | 0 | 0 | 0 | 5 | 5
  Hodgkin's Lymphoma | 0 | 2 | 0 | 5 | 7
  Non-Hodgkin's Lymphoma | 3 | 2 | 4 | 19 | 28
  Myelodysplastic Syndrome | 2 | 1 | 3 | 44 | 50
  Myeloproliferative Neoplasm | 0 | 0 | 0 | 5 | 5
  Other Acute Leukemia | 0 | 0 | 0 | 3 | 3
  Other Leukemia (including Chronic Lymphocytic Leukemia) | 0 | 1 | 0 | 2 | 3
  Severe Aplastic Anemia | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Engraftment With De-Escalating Umbilical Cord Total Nucleated Cell (TNC) Dose
Description: We aim to identify the lowest threshold of umbilical cord total nucleated cell (TNC) dose that can be utilized assure durable umbilical cord blood engraftment in the haplo-cord transplants. The threshold will be defined as the lowest dose which assures cord blood engraftment occurs in at least 80% of subjects.
Time Frame: 100 days
Population: A subset of participants were assessed to analyze the lowest threshold of umbilical cord total nucleated cell (TNC) dose. Once the lowest threshold was established, the remaining participants on study were treated based on that threshold.
Measure: Number; unit: participants
Groups:
- All Patients: Haplo-cord transplantation:
  For the transplant component of treatment, subject will receive umbilical cord blood. The study involves transplantation of unlicensed units of cord blood. Therefore, these are considered investigational products.
  In addition to the umbilical cord blood unit, recipients will receive stem cells from a family member ( a haplo-identical donor).
Arm/Group | All Patients
Number analyzed (Participants) | 60
participants
  Participants Achieving Engraftment with Minimum TNC of 2 x 10^5/kg: number analyzed (Participants) | 15
  Participants Achieving Engraftment with Minimum TNC of 2 x 10^5/kg | 15
  Participants Achieving Engraftment with Minimum TNC of 1 x 10^5/kg in umbilical cord blood unit: number analyzed (Participants) | 20
  Participants Achieving Engraftment with Minimum TNC of 1 x 10^5/kg in umbilical cord blood unit | 18
  Participants Achieving Engraftment with Minimum TNC of 0.5 x 10^5/kg: number analyzed (Participants) | 25
  Participants Achieving Engraftment with Minimum TNC of 0.5 x 10^5/kg | 20

2. Secondary Outcome: Long-term Survival of Subjects Undergoing Haplo-cord Transplants
Description: Evaluate the long term outcome of subjects undergoing haplo cord transplants using an optimally matched umbilical cord blood (UCB) graft (i.e. Survival, profession-free survival (PFS), Relapse, transplant-related mortality (TRM), toxicities, infections and GVHD)
Time Frame: 5 years after transplant
Reporting Status: Not Posted

3. Secondary Outcome: Impact of IPA Targeting on Transplant Outcome
Description: As much as possible, UCB units will be chosen to be IPA targeted. This is not always possible. We will therefore also retrospectively analyze transplant outcomes and correlate with IPA status.
Time Frame: 5 years from transplantation
Reporting Status: Not Posted

4. Secondary Outcome: Impact of NIMA Matching on Transplant Outcome
Description: As much as possible, UCB units will be chosen to be NIMA matched. This is not always possible. We will therefore also retrospectively analyze transplant outcomes and correlate with NIMA status.
Time Frame: 5 years from transplantation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all patients from start of transplant conditioning regimen through 1 year post-transplant or when the participant was removed from the study, whichever was sooner, assessed up to 1 year.
Description: Per protocol, events reported were grade 2 and higher infection and graft-versus-host disease events, and all other hematopoietic or extramedullary events grade 3 or higher per CTCAE v4.0.
Arm/Group | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg | Cohort 4
All-Cause Mortality (participants affected / at risk) | 6/15 | 6/20 | 11/25 | 79/210
Serious Adverse Events (participants affected / at risk) | 7/15 | 9/20 | 14/25 | 156/210
Other Adverse Events (participants affected / at risk) | 6/15 | 6/20 | 12/25 | 93/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg (N=15) | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg (N=20) | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg (N=25) | Cohort 4 (N=210)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious Colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Adenovirus Viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered Mental Status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders, other - Junctional rhythym (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cord blood unit clot (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cord colitis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cytomegalovirus meningoencephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus pneumonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cytomegalovirus Retinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus Viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 11 (11)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 11 (11)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Epstein-Barr Virus Viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Failure to Thrive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (11)
Fever (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fungal sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemolytic Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Herpes Simplex Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Human Herpes Virus 6 Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Infusion-related Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 5 (7) | 0 (0) | 0 (0) | 5 (7)
JC Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ Failure (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pericardial Tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 31 (33)
Post-operative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-transplant Lymphoproliferative Disorder (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 9 (9)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 5 (6) | 15 (16)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 21 (22)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sweet's Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxoplasmosis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Varicella zoster infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Veno-occlusive disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Graft-versus-Host Disease (Investigations) | 2 (2) | 0 (0) | 0 (0) | 18 (18)
Chronic Graft-versus-Host Disease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Graft Failure (Investigations) | 0 (0) | 0 (0) | 3 (3) | 10 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Minimum Cell Dose 2 x 10^7 TNC/kg (N=15) | Cohort 2 - Minimum Cell Dose 1 x 10^7 TNC/kg (N=20) | Cohort 3 - Minimum Cell Dose 0.5 x 10^7 TNC/kg (N=25) | Cohort 4 (N=210)
Cytomegalovirus viremia (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 30 (31)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
C. difficile colitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 30 (33)
Candida esophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Catheter Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B Reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human Herpes Virus 6 Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Herpes Simplex Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Infectious Diarrhea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 14 (14)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 11 (11)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vaginal yeast infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 9 (9)
Upper Respiratory Infection (Infections and infestations) | 4 (4) | 1 (1) | 5 (6) | 26 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT01810588/Prot_SAP_000.pdf